CLINICAL TRIAL: NCT06895668
Title: Self-harm and the Prison Environment (SHAPE): a Mixed Methods Study of the Role of Custody-specific Factors in Self-harm Behaviours Amongst Men and Women in Prison.
Brief Title: Self-harm and the Prison Environment Mixed Methods Study
Acronym: SHAPE
Status: Not yet recruiting | Type: Observational
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS350490; NIHR304724 (Other Grant/Funding Number: NIHR)
Record Dates: First submitted 2025-03-17; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Self-Harm; Self-harm Behavior; Self-Harm, Deliberate
Keywords: Self-harm; Self-injury; Prospective cohort study; Qualitative; Focus groups; Semi-structured interviews; Environmental factors; Prison; Custody; Offenders; Prisoners; Incarceration
MeSH Terms: conditions — Self-Injurious Behavior | interventions — Cohort Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Prison entry cohort: Cohort of 458 prisoners from two men's local (remand) prisons and one female high security prison in England, recruited on entry to prison using series of random samples of prison admissions across the recruitment period.
  Interventions: Other: None (cohort study)

INTERVENTIONS:
Other: None (cohort study) — None (cohort study)

SUMMARY:
Self-harming behaviour is a major problem in UK prisons: the number of self-harm incidents has more than doubled over the past decade. People who self-harm in prison are at greater risk of subsequent death by suicide. Risk assessment processes for the prison population are rudimentary and critically under-informed. Research evidence shows that a person's life history and current mental health make some more vulnerable than others to such behaviour. However, the role of the prison environment in contributing to self-harm risk is poorly understood. A wide range of environmental factors might be important, such as the degree of contact with the outside world, stimulation in the daily regime and conflicts with peers and prison staff. In a pilot study that the investigators carried out in a male prison, prison environment characteristics such as placement in a single-occupancy cell and changing cell or cellmate more frequently were associated with self-harm. These environmental factors now require further study in larger-scale research in men and women's prisons. Understanding which environmental factors are relevant to self-harming behaviour will help prison and healthcare staff to make better informed assessments of self-harming risks and better management plans to reduce such behaviours.

This study aims to establish the impact of the prison environment on self-harming behaviour amongst both men and women in prison using a mixed methods approach. The investigators now want to establish the precise influence of such factors in both male and female prisoners to help to improve the management of such behaviour. This will be done by interviewing and following up groups of male and female prisoners for a 12 week period (the cohort study). The investigators will then use focus groups to explore prisoner, staff and other stakeholder views on the findings (the focus group study). Finally, female self-harming prisoners will be interviewed to explore the detailed perspectives of women (the interview study). The studies will take place at three prisons: HMP Wandsworth and HMP Pentonville (both medium security men's prisons) and HMP Bronzefield (a high security women's prison).

Cohort study: Adults entering either prison are eligible to participate. The investigators will recruit a random sample of 458 men and women (based on a power calculation informed by previous pilot work). Participants will complete two 1-hour baseline assessments before being followed up for 12 weeks. The researchers will conduct two further in-person assessments and examine the participant's health and custodial records at the prison and link this with local wing-level prison data. The results will establish which of a range of possible prison environmental factors are related to self-harming behaviour.

The following prison-related predictors of self-harm behaviour will be examined in the cohort study:

* Placement in a single-occupancy cell
* Frequency of cell changes
* Placement in solitary confinement
* Violence perpetration
* Other disciplinary infractions
* Violent/sexual victimisation
* Work status in prison
* Time in purposeful activities
* Social visit status
* Legal status
* Time out of cell (cumulative exposure)
* Staffing ratio (cumulative exposure)
* Staff experience (cumulative exposure)
* Staff responsivity to emergency bells (cumulative exposure)

Focus group study: The researchers will then use focus groups to explore the perspectives of prisoners and staff on our research findings and their implications for day-to-day practice. Adult self-harming prisoners, peer support workers, supervising officers and healthcare staff at the same prisons, alongside other stakeholders working in the field - including carers - will be eligible to participate in audio-recorded focus groups.

Interview study: The investigators will explore in more detail the impact of prison-related factors on self-harm behaviour amongst female prisoners (having already completed such interviews with male prisoners in our pilot work). 10 adult self-harming women at HMP Bronzefield will be recruited to take part in audio-recorded semi-structured interviews.

Answering these questions will help to inform prison-wide strategies for reducing self-harm in both male and female prisoners.

ELIGIBILITY:
Inclusion Criteria:

- New entrants to prison

Exclusion Criteria:

* Expected release/transfer date less than 12 weeks from date of entry
* Lack capacity to give informed consent
* Insufficient spoken English skills to participate
* Assessed persistently as not safe to be seen face to face due to imminent high risk of violence.
* Risk of psychological harm from participation more than minimal (based on risk assessment with prison's Safer Custody and mental health teams)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People entering one of three prisons in England
Sampling Method: Probability Sample
Enrollment: 458 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Self-harm behaviour | From enrolment to the end of observation at 12 weeks
  Self-harm behaviour (any) in time-to-event format, assessed using a modified version of the Columbia - Suicide Severity Rating Scale (C-SSRS). Outcome will be self-harm behaviour survival time, analysed using a survival analysis approach (Cox shared frailty modelling) to produce Hazard Ratios for each predictor.

SECONDARY OUTCOMES:
Suicidal ideation | From enrollment to the end of observation at 12 weeks
  Suicidal ideation (any) in binary format, assessed using a modified version of the Columbia - Suicide Severity Rating Scale (C-SSRS).